CLINICAL TRIAL: NCT06080425
Title: Addressing Intergenerational Obesity and Promoting Healthy Eating and Physical Activity Among Individuals [PIHRK'D] Living With Diabetes in Rural Kentucky
Brief Title: Promoting Intergenerational Health in Rural Kentuckians With Diabetes (PIHRK'D)
Acronym: PIHRK'D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-0225; 3048115811 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Monthly in-home MNT will be conducted by the RD for members of the household but will be tailored for the participant with diabetes for 6 months. Dietary counseling will be focused on living with diabetes, appropriate food choices, glycemic control, and importance of weight management. To enhance participant buy-in and sustainability, the RD will utilize Motivational Interviewing (MI) principles to work with participants to improve self-efficacy of behavior change and set Specific, Measurable, Achievable, Relevant, and Time-Bound (SMART) goals each month.
  Also, participants will enroll in the group facilitated Dining with Diabetes program with the option to bring one member of their social to their local Cooperative Extension offices. Dining with Diabetes is an interactive 4-session program that includes direct education on healthy eating, food preparation strategies, physical activity, emotional health, identifying complications of diabetes, and problem-solving skills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Nutrition Therapy (Other): Medical Nutrition therapy is an intervention that will be administered to the participants for 6 months.
  Interventions: Behavioral: Medical Nutrition Therapy

INTERVENTIONS:
Behavioral: Medical Nutrition Therapy — Counselling

SUMMARY:
The goal of this feasibility study is to use family units as support to promote nutrition and physical activity of individuals with type 2 diabetes. The main question it aims to answer is:

• How does the family structure impact the health of its members living with type 2 diabetes?

Participants will be asked to;

* Tell us about their access to food sources and places in the community to engage in physical activity.
* A nutrition and physical activity plan will be developed for participants and their families to use for 6 months.

DETAILED DESCRIPTION:
The proposed project is informed by the National Framework for Health Equity and Well Being, which was recently developed by the Cooperative Extension Service. This framework explicitly acknowledges the multiple levels of influence on health outcomes and the role of Cooperative Extension Service as a mitigator of community-level health inequities. The framework acknowledges factors that contribute to health inequities at various societal levels, including root causes of structural inequity; norms, policies, and practices; and social determinants of health. As individuals flow through multiple sectors of the environment, each is known to have a direct influence individually and collectively. For the proposed grant, the study will focus on how county-level Extension agents (federally funded program) can be used to mitigate health disparities that contribute to intergenerational obesity and T2DM management in rural Kentucky. Community-level factors also impact health outcomes, such as lack of access to healthy, affordable food, as well as availability of health-related resources. Community assets will be gathered using subjective and objective community audits and assessed at the participant level using social network analysis. Societal-level factors include social norms and cultural health beliefs that impact health decision-making within the community, particularly families/households.

Participants will be recruited on a staggered basis from 2 rural counties in Kentucky. Recruitment will be conducted via Extension Offices, word-of-mouth, social media, UK Healthcare outpatient clinics (e.g., internal medicine, family medicine, endocrinology), as well as UK's Barnstable Brown Diabetes and Obesity Center. Once enrolled, participants will be screened by the RD to confirm obesity/overweight, T2DM diagnosis, and identify each participant's placement within the Transtheoretical Model (Six Stages of Change): pre-contemplation, contemplation, preparation, action, maintenance, or relapse. The enrollment stage of change will be used to develop appropriate goals for each participant. Beyond the primary enrolled participant in the study, members of the household will be invited to attend meetings with the RD and Dining with Diabetes program sessions.

Aim 1: Use social network analysis to describe (a) community assets (e.g., access to healthy eating and ways to participate in physical activity) and (b) intergenerational links to obesity and diabetes (e.g., parent, sibling, child).

Social network analysis will be used to map food sources and food assistance (e.g., supermarket, convenience store, fast food, food pantries), including the types of food offered and frequency of engagement with food sources. Similar methods will be used to identify areas/places within the community that could be used to engage in physical activities (e.g., gym, community center, green space, walking trails). A network map will be developed per household to be used to develop a tailored program that that is feasible and accessible to overweight/obese individuals living with diabetes and members of their household.

Participants will be asked to provide the following information on up to 5 immediate family members: age; sex; education level; relationship (e.g., spouse, child, sibling, parent); whether that individual is overweight/obese; and current T2DM diagnosis status (e.g., no diagnosis, diagnosed by a healthcare provider, told by a healthcare provider to be prediabetic). Additional information will be gathered regarding the interconnectedness (e.g., person 1 and person 3 are siblings) of the known relationships between family members.

Aim 2: Develop a household-specific nutrition and physical activity plan. A 6-month nutrition and physical activity intervention will be implemented with eligible, enrolled Kentucky residents focused on leveraging household/familial social networks. Medical nutrition therapy will be used within a household to tailor healthy eating and physical activity. The 4-week Dining with Diabetes Program will be used to supplement medical nutrition therapy. The participant will be engaged to take someone from their household with them to the Dining with Diabetes sessions to promote and reinforce healthy lifestyle choices.

At the baseline study visit, the research coordinator will provide a study overview and conduct consent. After consent has been obtained, the research coordinator will collect demographics, baseline clinical outcomes, validated surveys, and social network data for the perceived community resources and family characteristics. The research coordinator will conduct an objective community assessment and provide that information as well as the perceived community assets data to the dietitian to be used as part of the medical nutrition therapy. The research coordinator will collect relevant clinical measures, specifically blood pressure, HbA1c, and lipid panel, and validated surveys at baseline and 3 and 6 months post-intervention. The dietitian will schedule and complete the first session medical nutrition therapy within 2 weeks of baseline data collection and will continue to conduct medical nutrition therapy monthly for 6 months. The dietitian will also collect relevant clinical measures, specifically blood pressure, HbA1c, and lipid panel, and validated surveys at 3 and 6 months during the intervention period.

Aim 3: Determine the preliminary effectiveness of tailored nutrition and physical activity for those living within the household.

Data will be collected at five times per participant throughout the intervention. Data collection time points will include baseline and twice during the 6 months intervention period (3 and 6 months) and then again at 3 months and 6 months post-intervention.

To evaluate the feasibility of the proposed intervention, the investigators will use guiding questions that address the following: evaluation of recruitment capability and resulting sample characteristics, evaluation and refinement of data collection procedures and outcome measures, evaluation of acceptability and suitability of intervention and study procedures, evaluation of resources and ability to manage and implement the study and intervention, and preliminary evaluation of participant responses to interventions. Acceptability of community health workers will be assessed using a previously published assessment of community health workers. This assessment measures attributes, such as the participants' perception of cooperative extension agents and a registered dietician to address health concerns, respect and dignity, honesty, interpersonal relationships, and assistance with changing behaviors.

ELIGIBILITY:
Inclusion Criteria:

* must be diagnosed with type 2 diabetes
* must be from rural Kentucky
* must be living in rural Kentucky for at least 1 year

Exclusion Criteria:

* potential participants without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
hemoglobin A1c values measured at the five post-baseline follow-up points | baseline, 3 months, 6 months, 9 months and 12 months
  This is a test that measures average blood sugar levels over the past 3 months
body weight measured at the five post-baseline follow-up points | baseline, 3 months, 6 months, 9 months and 12 months
  This is an indices used in the estimation of BMI

SECONDARY OUTCOMES:
Diabetes Knowledge | baseline, 3 months, 6 months, 9 months and 12 months
  Diabetes knowledge of the participants will be assessed using a validated Diabetes Knowledge Questionnaire (DKQ). The DKQ is a 24-item questionnaire, designed by Starr County Diabetes Education Study, to elicit information about patients' understanding of the cause of their disease, its associated complications, blood glucose levels, diet, and physical activity. The DKQ has three response options "yes", "no", and "don't know". One point is awarded for each correct option, whereas, no point or negative scoring for the incorrect option. Its scoring involves summing-up the points obtained by each participant. A higher score represents better disease knowledge.
Diabetes self-management | baseline, 3 months, 6 months, 9 months and 12 months
  Diabetes self-management/self-efficacy will be assessed using the Diabetes Empowerment Scale. Diabetes Empowerment Scale is a 28-item scale that measures diabetes-related psychosocial self-efficacy with an overall Cronbach's uses 3 subscales: Managing the Psychosocial Aspects of Diabetes, Assessing Dissatisfaction and Readiness to Change, and Setting and Achieving Diabetes Goals (Anderson et al, 2000).
  The questionnaires consist of 28 items with 3 subscales, with each item rated along a 5-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree). The range of score is divided in three subgroups as low (28-65 scores), middle (66-103) and high (104-140).
Dietary Intake | baseline, 3 months, 6 months, 9 months and 12 months
  24-hour dietary will be used to estimate the dietary intake of the participants
Diabetes Distress | baseline, 3 months, 6 months, 9 months and 12 months
  The Diabetes Distress Scale (DDS) is a 17-item scale that measures patient concerns about disease management, support, emotional burden and access to care. The response scale for each question ranges from "1" (not a problem) to "6" (a very serious problem). An average score of greater than or equal to 3 indicated moderate distress and discriminated between high and low distressed groups (Fisher et al, 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Smalls, PhD, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The participants have been informed that their personal data will not be shared, and their confidentiality will be kept.

REFERENCES:
- [Result] Albuquerque D, Nobrega C, Manco L, Padez C. The contribution of genetics and environment to obesity. Br Med Bull. 2017 Sep 1;123(1):159-173. doi: 10.1093/bmb/ldx022. PMID 28910990
- [Result] Ali O. Genetics of type 2 diabetes. World J Diabetes. 2013 Aug 15;4(4):114-23. doi: 10.4239/wjd.v4.i4.114. PMID 23961321
- [Result] Anders S, Schroeter C. Diabetes, diet-health behavior, and obesity. Front Endocrinol (Lausanne). 2015 Mar 16;6:33. doi: 10.3389/fendo.2015.00033. eCollection 2015. PMID 25852643
- [Result] Anderson RM, Funnell MM, Fitzgerald JT, Marrero DG. The Diabetes Empowerment Scale: a measure of psychosocial self-efficacy. Diabetes Care. 2000 Jun;23(6):739-43. doi: 10.2337/diacare.23.6.739. PMID 10840988
- [Result] Baig AA, Benitez A, Quinn MT, Burnet DL. Family interventions to improve diabetes outcomes for adults. Ann N Y Acad Sci. 2015 Sep;1353(1):89-112. doi: 10.1111/nyas.12844. Epub 2015 Aug 6. PMID 26250784
- [Result] Benjamini Y., Hochberg Y. (1995). Controlling the False Discovery Rate: A Practical and Powerful Approach to Multiple Testing. Journal of the Royal Statistical Society. Series B (Methodological), 57(1), 289-300
- [Result] Bhupathiraju SN, Hu FB. Epidemiology of Obesity and Diabetes and Their Cardiovascular Complications. Circ Res. 2016 May 27;118(11):1723-35. doi: 10.1161/CIRCRESAHA.115.306825. PMID 27230638
- [Result] Chapman-Novakofski K, Karduck J. Improvement in knowledge, social cognitive theory variables, and movement through stages of change after a community-based diabetes education program. J Am Diet Assoc. 2005 Oct;105(10):1613-6. doi: 10.1016/j.jada.2005.07.010. PMID 16183364
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Result] Demir D, Bektas M. The effect of childrens' eating behaviors and parental feeding style on childhood obesity. Eat Behav. 2017 Aug;26:137-142. doi: 10.1016/j.eatbeh.2017.03.004. Epub 2017 Mar 22. PMID 28363115
- [Result] Fisher L, Glasgow RE, Mullan JT, Skaff MM, Polonsky WH. Development of a brief diabetes distress screening instrument. Ann Fam Med. 2008 May-Jun;6(3):246-52. doi: 10.1370/afm.842. PMID 18474888
- [Result] Fruh SM. Obesity: Risk factors, complications, and strategies for sustainable long-term weight management. J Am Assoc Nurse Pract. 2017 Oct;29(S1):S3-S14. doi: 10.1002/2327-6924.12510. PMID 29024553
- [Result] Garcia AA, Villagomez ET, Brown SA, Kouzekanani K, Hanis CL. The Starr County Diabetes Education Study: development of the Spanish-language diabetes knowledge questionnaire. Diabetes Care. 2001 Jan;24(1):16-21. doi: 10.2337/diacare.24.1.16. PMID 11194219
- [Result] Griffie D, James L, Goetz S, Balotti B, Shr YH, Corbin M, Kelsey TW. Outcomes and Economic Benefits of Penn State Extension's Dining With Diabetes Program. Prev Chronic Dis. 2018 May 3;15:E50. doi: 10.5888/pcd15.170407. PMID 29729134
- [Result] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284
- [Result] Hood KK, Hilliard M, Piatt G, Ievers-Landis CE. Effective strategies for encouraging behavior change in people with diabetes. Diabetes Manag (Lond). 2015;5(6):499-510. PMID 30100925
- [Result] Hoogland AI, Hoogland CE, Bardach SH, Tarasenko YN, Schoenberg NE. Health Behaviors in Rural Appalachia. South Med J. 2019 Aug;112(8):444-449. doi: 10.14423/SMJ.0000000000001008. PMID 31375842
- [Result] Kirkman MS, Briscoe VJ, Clark N, Florez H, Haas LB, Halter JB, Huang ES, Korytkowski MT, Munshi MN, Odegard PS, Pratley RE, Swift CS. Diabetes in older adults. Diabetes Care. 2012 Dec;35(12):2650-64. doi: 10.2337/dc12-1801. Epub 2012 Oct 25. No abstract available. PMID 23100048
- [Result] Kritchevsky SB. Taking Obesity in Older Adults Seriously. J Gerontol A Biol Sci Med Sci. 2017 Dec 12;73(1):57-58. doi: 10.1093/gerona/glx228. No abstract available. PMID 29240912
- [Result] Lawrence JM, Divers J, Isom S, Saydah S, Imperatore G, Pihoker C, Marcovina SM, Mayer-Davis EJ, Hamman RF, Dolan L, Dabelea D, Pettitt DJ, Liese AD; SEARCH for Diabetes in Youth Study Group. Trends in Prevalence of Type 1 and Type 2 Diabetes in Children and Adolescents in the US, 2001-2017. JAMA. 2021 Aug 24;326(8):717-727. doi: 10.1001/jama.2021.11165. PMID 34427600
- [Result] Martire LM, Helgeson VS. Close relationships and the management of chronic illness: Associations and interventions. Am Psychol. 2017 Sep;72(6):601-612. doi: 10.1037/amp0000066. PMID 28880106
- [Result] Massey, C.N., Appel, S.J., Buchanan, K.L., et al. (2010) Improving Diabetes Care in Rural Communities: An Overview of Current Initiatives and a Call for Renewed Efforts. Clinical Diabetes, 28, 20-27. http://dx.doi.org/10.2337/diaclin.28.1.20
- [Result] Mayberry LS, Berg CA, Greevy RA Jr, Wallston KA. Assessing helpful and harmful family and friend involvement in adults' type 2 diabetes self-management. Patient Educ Couns. 2019 Jul;102(7):1380-1388. doi: 10.1016/j.pec.2019.02.027. Epub 2019 Mar 1. PMID 30922622
- [Result] Misra R, Fitch C. A model exploring the relationship between nutrition knowledge, behavior, diabetes self-management and outcomes from the dining with diabetes program. Prev Med. 2020 Dec;141:106296. doi: 10.1016/j.ypmed.2020.106296. Epub 2020 Oct 23. PMID 33132185
- [Result] Okobi OE, Ajayi OO, Okobi TJ, Anaya IC, Fasehun OO, Diala CS, Evbayekha EO, Ajibowo AO, Olateju IV, Ekabua JJ, Nkongho MB, Amanze IO, Taiwo A, Okorare O, Ojinnaka US, Ogbeifun OE, Chukwuma N, Nebuwa EJ, Omole JA, Udoete IO, Okobi RK. The Burden of Obesity in the Rural Adult Population of America. Cureus. 2021 Jun 20;13(6):e15770. doi: 10.7759/cureus.15770. eCollection 2021 Jun. PMID 34295580
- [Result] Rollnick S, Butler CC, Kinnersley P, Gregory J, Mash B. Motivational interviewing. BMJ. 2010 Apr 27;340:c1900. doi: 10.1136/bmj.c1900. No abstract available. PMID 20423957
- [Result] Schmitt A, Gahr A, Hermanns N, Kulzer B, Huber J, Haak T. The Diabetes Self-Management Questionnaire (DSMQ): development and evaluation of an instrument to assess diabetes self-care activities associated with glycaemic control. Health Qual Life Outcomes. 2013 Aug 13;11:138. doi: 10.1186/1477-7525-11-138. PMID 23937988
- [Result] Schor EL. The influence of families on child health. Family behaviors and child outcomes. Pediatr Clin North Am. 1995 Feb;42(1):89-102. doi: 10.1016/s0031-3955(16)38910-6. PMID 7854880
- [Result] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Result] Strasser B. Physical activity in obesity and metabolic syndrome. Ann N Y Acad Sci. 2013 Apr;1281(1):141-59. doi: 10.1111/j.1749-6632.2012.06785.x. Epub 2012 Nov 21. PMID 23167451
- [Result] Swift DL, Johannsen NM, Lavie CJ, Earnest CP, Church TS. The role of exercise and physical activity in weight loss and maintenance. Prog Cardiovasc Dis. 2014 Jan-Feb;56(4):441-7. doi: 10.1016/j.pcad.2013.09.012. Epub 2013 Oct 11. PMID 24438736
- [Result] van Dijk SJ, Molloy PL, Varinli H, Morrison JL, Muhlhausler BS; Members of EpiSCOPE. Epigenetics and human obesity. Int J Obes (Lond). 2015 Jan;39(1):85-97. doi: 10.1038/ijo.2014.34. Epub 2014 Feb 25. PMID 24566855
- [Result] Weihs, K., Fisher, L., & Baird, M. (2002). Families, health, and behavior: A section of the commissioned report by the Committee on Health and Behavior: Research, Practice, and Policy Division of Neuroscience and Behavioral Health and Division of Health Promotion and Disease Prevention Institute of Medicine, National Academy of Sciences. Families, Systems, & Health, 20(1), 7-46. https://doi.org/10.1037/h0089481
- [Derived] Smalls BL, Ortz CL, Barr-Porter M, Norman-Burgdolf H, McLouth CJ, Harlow B, Leshi O. Promoting Intergenerational Health in Rural Kentuckians With Diabetes (PIHRK'D): Protocol for a Longitudinal Cohort Study. JMIR Res Protoc. 2025 Jul 24;14:e69301. doi: 10.2196/69301. PMID 40705414
- See also: National Institute for Diabetes and Digestive and Kidney Diseases. (2016). Diabetes diet, eating, and physical activity — https://www.niddk.nih.gov/health-information/diabetes/overview/diet-eating-physical-activity
- See also: State of Childhood Obesity. Kentucky Rates. 2020 — https://stateofchildhoodobesity.org/state-data/?state=ky